CLINICAL TRIAL: NCT04483050
Title: The Clinical Effect of Hip Protection Orthosis for the Hip Protection of Hip Dislocation in Patients With Severe Neuromuscular Disease, Open Label, Pilot Study
Brief Title: The Clinical Effect of Hip Protection Orthosis for the Hip Protection of Hip Dislocation in Patients With Severe Neuromuscular Disease, Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-2002/594-305
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Device: Hip protection orthosis

INTERVENTIONS:
Device: Hip protection orthosis — Experimental group would wear hip protection orthosis over 12 hours a day for 1 year.

SUMMARY:
The Clinical Effect of Hip Protection Orthosis for the Hip Protection of Hip Dislocation in Patients With Severe Neuromuscular Disease

ELIGIBILITY:
Inclusion Criteria:

* age from 1 to 15
* Patients with severe neuromuscular disease
* Patients who agreed to participate in the study
* Hip dislocation more than 10% (migration index)

Exclusion Criteria:

* If do not agree with the study
* Those who are determined to be difficult to participate under the judgment of the research director
* History of hip joint surgery

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Migration index | 6 months
  Hip AP radiography

SECONDARY OUTCOMES:
Cobb's angle (') | 6 months
  using radiography, expressed by degree from 0' to 180'. The closer to 0', the better the value.
Range of motion of hip joint (') | 6 months
  Using goniometer, measure the hip and knee abduction and flexion angle expressed by degree from 0' to 180'. The closer to 180', the better the value.
Visual analog scale | 6 months
  measure the pain expressed by score from 0 to 10. The closer to 10, the higher the pain.
Likert scale (score) | immediately after wearing orthosis
  measure the satisfaction about hip protection orthosis expressed by score from 0 to 5. The closer to 5, the higher the satisfaction.
Child Health Index of Life with Disabilities (CPCHILD) | 6 months
  measure the quality of life expressed by score from 0 to 100. The higher the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Juseok Ryu, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, Seongnam-si, Gyeonggi-do, South Korea